CLINICAL TRIAL: NCT07133451
Title: Prospective Cohort Registry Study on Multimodal Imaging Evaluation of Vulnerability of Intracranial and Extracranial Atherosclerotic Plaques: A Comparison of HR-VWI, OCT, and RWS
Brief Title: Multimodal Imaging Evaluation of Vulnerability of Atherosclerotic Plaques: A Comparison of HR-VWI, OCT, and RWS
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai Jiao Tong University Affiliated Sixth People's Hospital (Other)
Responsible Party: Principal Investigator, Yueqi Zhu, Professor, Shanghai Jiao Tong University Affiliated Sixth People's Hospital
Other Study IDs: Plaque-MAGIC Study
Record Dates: First submitted 2025-08-06; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Intracranial Atherosclerotic Stenosis
Keywords: high resolution magnetic resonance imaging; intracranial atherosclerotic stenosis; atherosclerotic Plaques; radial Wall Strain; optical Coherence Tomography
MeSH Terms: conditions — Plaque, Atherosclerotic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with moderate to severe stenosis (stenosis degree: 70% ~ 99%) in both intracranial and extr: Patients with moderate to severe stenosis (stenosis degree: 70% ~ 99%) in both intracranial and extracranial arteries were considered for enrollment in this study.

SUMMARY:
The primary objective of this study is to evaluate the vulnerability of intracranial and extracranial atherosclerotic plaques using HR-VWI, OCT, and RWS technologies, while exploring correlations among these three imaging techniques. Secondary objectives include: 1) Investigating the relationship between RWS and plaque progression and identifying optimal RWS predictors; 2) Further evaluating the clinical value of RWS and HR-VWI in stroke prediction through two-year clinical and HR-VWI follow-up evaluations.

DETAILED DESCRIPTION:
Intracranial atherosclerotic stenosis (ICAS) is one of the leading causes of ischemic cerebrovascular disease worldwide, with an incidence rate as high as 46.6% among ischemic stroke or transient ischemic attacks (TIA) patients in China. Traditional arterial imaging techniques such as computed tomography angiography (CTA), magnetic resonance angiography (MRA), and digital subtraction angiography (DSA) all provide lumen imaging capabilities. However, these methods can only reflect the severity of atherosclerotic lesions through vascular narrowing, failing to accurately assess the condition of the vessel wall.

High resolution magnetic resonance vessel wall imaging (HR-VWI) has enabled 2D and 3D imaging of intracranial arterial walls. This technique not only provides clear visualization of vascular morphology and signal characteristics, but also identifies plaque components, enhancement intensity, reconstruction type and load by suppressing intravascular blood flow. It also evaluates ICAS-prone plaque features such as intraplaque hemorrhage (IPH), lipid-rich necrotic core (LRNC), and others. However, current HR-VWI scans face challenges including prolonged examination time, difficulties in aligning multiple sequences, and numerous contraindications (e.g., claustrophobia and pacemaker implantation). Additionally, image quality and effectiveness of intracranial artery HR-VWI are influenced by hardware/software parameters like magnetic field strength, receiving coils, imaging dimensions, sequences, and spatial resolution. These factors lead to variations across hospitals, with the absence of standardized protocols hindering standardized interpretation and analysis of images.

Optical Coherence Tomography (OCT), as an intravascular imaging technique, demonstrates high sensitivity and specificity in identifying different plaque components. With image resolution reaching 10μm - ten times that of conventional intravascular ultrasound- it has gained widespread recognition in coronary artery diagnosis and treatment. In recent years, OCT has also been applied in cerebral vascular interventional therapy, achieving notable progress in evaluating cerebral atherosclerotic plaques, performing interventional procedures, and conducting long-term follow-up studies.

Blood vessels are constantly subjected to biomechanical forces in the human body, including intraluminal arterial pressure and blood flow resistance. These mechanical forces induce dynamic strain and stress on vascular walls, which can trigger the rupture of atherosclerotic fibrous caps and inflammatory-prone plaques. High-resolution angiography can capture plaque strain or stress. Radial Wall Strain (RWS), a novel technique that utilizes high-resolution angiographic images and artificial intelligence to calculate plaque strain based on deformation patterns during different cardiac phases, has proven effective in coronary artery research. It demonstrates significant potential for risk stratification and prognosis prediction. Validation studies using OCT-defined plaque characteristics revealed that RWSmax shows a significant positive correlation with plaque lipid load and the lipid-fibrous cap ratio, while showing a significant negative correlation with cap thickness. A clinical cohort study employing propensity score matching evaluated the predictive power of angiography-based RWS for acute myocardial infarction (AMI) risk in newly diagnosed patients with mild-to-moderate coronary stenosis. Results indicated that RWSmax> 12% significantly increased the risk of AMI in untreated lesions by 7.25. Another study analyzed 1,318 delayed revascularization (DRV) vessels reported in the FAVOR III China main study. Vessels with RWSmax> 12% showed a 1-year vascular-derived composite endpoint event risk of 14.3%, compared to 2.9% for those ≤12% (risk ratio: 4.44). The research supports applying the novel RWS technology to assess residual risk in non-ischemic vessels defined by quantitative flow ratio (QFR), guiding necessary interventions such as intensified pharmacotherapy to enhance DRV safety. These findings indicate that RWS offers a novel decision-making model for coronary risk assessment and optimized management. Importantly, RWS can be calculated using routine single-slice angiographic images, eliminating the need for additional invasive procedures and demonstrating broad clinical applicability. However, its value in evaluating intracranial unstable plaques and their progression remains unverified. To address these technical advantages, this prospective clinical study aims to investigate RWS's efficacy in assessing intracranial plaque stability and progression risks, while comparing it with OCT and HR-VWI methods to evaluate feasibility and effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old;
* Severe stenosis of intracranial arteries (stenosis degree: 70% ~ 99%, traditional angiography is required to confirm the degree of stenosis according to the criteria of Warfarin-Aspirin Symptomatic Intracranial Disease (WASID) study);
* Carry out cerebral angiography and OCT within one week after HR-VWI examination;
* The patient or the legal representative of the patient is able and willing to sign an informed consent form.

Exclusion Criteria:

* Non-atherosclerotic intracranial and extracranial artery stenosis, such as dissection, smoke disease, etc.;
* There are contraindications to MRI, such as claustrophobia, metal implants, etc.; Renal insufficiency, elevated serum creatinine (more than twice the upper limit of normal);
* Patients with severe cardiopulmonary diseases were considered unsuitable for this study;
* Allergy to iodine or gadolinium contrast agent;
* Participants who were unable to complete the study due to mental illness, cognitive or emotional disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with moderate to severe stenosis (stenosis degree: 70% ~ 99%) in both intracranial and extracranial arteries were considered for enrollment in this study.
Sampling Method: Non-Probability Sample
Enrollment: 561 (Estimated)
Dates: Start 2025-08-10 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Diameter stenosis rate | 2024.8-2027.12
  According to the 3D TOF-MRA measurement of the lumen diameter at the narrowest part of the intracranial artery and the normal lumen diameter at the proximal end of the stenosis, the stenosis rate was calculated according to the WASID standard: diameter stenosis rate = [1- (the diameter at the narrowest part / the normal diameter at the proximal end of the stenosis)] × 100%
Identify different plaque components | 2024.8-2027.12
OCT scanning scheme and image analysis | 2024.8-2027.12
  This study utilized the ILUMIEN OPTIS system (Abbott Medical, USA) to obtain frequency-domain OCT (FD-OCT) images. The procedure was performed under general anesthesia. Patients first underwent DSA cerebral angiography, after which a 6F long sheath (Epsylar, Opti Med, USA) was placed proximal to the lesion. A distal access catheter was introduced near the target lesion, and under fluoroscopy guidance, a micro guidewire was advanced through the lesion into the normal arterial lumen distally. The Dragonfly OPTIS imaging catheter (Abbott Medical, USA) was then exchanged for standard "single-track" entry, guiding it into the target vascular lesion. A mixed solution of physiological saline and iohexol contrast agent (GE Healthcare, Cork, Ireland), with a 1:1 concentration, was injected via the distal access catheter. OCT images were captured using automated retraction technology during blood clearance.
RWS | 2024.8-2027.12
  Using single-position angiographic sequences, the cardiac cycle inference algorithm and automatic frame selection algorithm were applied to identify a key frame and multiple analysis frames with high image quality distributed across different phases of the same cardiac cycle. Subsequently, vascular segments of interest were defined on the key frame, and all corresponding matching segments were obtained through keypoint matching algorithms. The sub-pixel vascular contour segmentation algorithm was then used to generate detailed vessel outlines and calculate radial diameters for all analysis frames. Based on multi-frame vascular contours and diameter data, an automatic 2D point cloud registration algorithm was employed to determine radial alignment relationships between vascular segments. Finally, relative radial deformation was calculated using these alignment relationships and diameter information to derive RWS variation curves.

CONTACTS AND LOCATIONS:
Overall Officials: Yueqi Zhu, MD, Principal Investigator — Shanghai Jiao Tong University Affiliated Sixth People's Hospital
Locations (1):
- Shanghai 6th People's Hospital, Shanghai, China